CLINICAL TRIAL: NCT02579200
Title: Inspiratory Muscle Training for Dyspneic Patients With COPD-HF Overlap: a Multicenter, Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training for Breathless Patients With Chronic Obstructive Pulmonary Disease and Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Collaborators: KU Leuven (Other); Federal University of São Paulo (Other); Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Dr. J. Alberto Neder, Study Chair, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT COPD+HF
Record Dates: First submitted 2015-03-10; First posted 2015-10-19 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Heart Failure, Systolic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiratory Muscle Training (IMT) (Active Comparator): POWERbreathe®KHA (IMT group)
  Interventions: Device: POWERbreathe®KHA (IMT group)
- Sham Training (Sham Comparator): POWERbreathe®KH2 (sham group)
  Interventions: Device: POWERbreathe®KH2 (sham group)

INTERVENTIONS:
Device: POWERbreathe®KHA (IMT group) — 2 training sessions/day consisting of 30 breaths (~50% maximal inspiratory pressure; Pi,max), 7 days/week (once/week supervised at research center), for 8 weeks using an electronic tapered flow resistive loading (TFRL) device (POWERbreathe®KH2, HaB International Ltd., Southam, UK). Measurements of PImax will be performed every week and training loads will be increased continuously to maintain the actual ~50% Pimax values.
  Arms: Inspiratory Muscle Training (IMT)
Device: POWERbreathe®KH2 (sham group) — 2 training sessions/day of 30 breaths at an inspiratory load of no more than 10% of their initial Pi,max (POWERbreathe®KH2, HaB International Ltd., Southam, UK). This training load will not be changed during the entire study period.
  Arms: Sham Training

SUMMARY:
The purpose of this study is to determine whether inspiratory muscle training is effective to improve breathless and exercise intolerance in symptomatic patients with chronic obstructive pulmonary disease (COPD) plus chronic heart failure (HF).

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) and heart failure with reduced left ventricular ejection fraction (HF) are leading causes of disability and death worldwide. Unfortunately, COPD and HF coexist in up to a third of elderly patients making the so-called COPD-HF overlap (CHO) a major challenge to Health Care Systems. In addition, population ageing anticipates that CHO prevalence will further increase in the next decades.

Intolerance to exertion due to disabling breathlessness is the hallmark of COPD and HF and these abnormalities are notoriously potentiated by diseases coexistence.

The inspiratory muscles are centrally related to the pathophysiology of exertional dyspnea in COPD and HF. In both populations a higher central motor command output is required to maintain adequate force generation in the face of weaker inspiratory muscles. This information is interpreted as "shortness of breath".

There is well established evidence gained from recent meta-analyses indicating that inspiratory muscle training (IMT), as a standalone therapy, significantly improves inspiratory muscle function (strength and endurance), dyspnea during daily activities, and functional exercise capacity in COPD and HF. Previous findings indicate that reduced pressure-generating capacity reflecting inspiratory muscle weakness is frequently observed in patients with COPD-HF and related to a clinically-relevant outcome: exertional dyspnea. These findings set the scene for a randomized controlled trial to investigate the potential role of IMT in dyspnea palliation in CHO patients.

Objectives

To determine the effects of IMT on:

1. Dyspnea on daily life
2. Inspiratory muscle strength and endurance
3. Dyspnea on exertion and time to exercise intolerance

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnoses of COPD and HF under optimized clinical treatment as judged by the accompanying physician
* Reduced left ventricular ejection fraction (<50%)
* Non-reversible airway obstruction (post-bronchodilator FEV1/FVC < 0.7 and FEV1 < 80 %)
* Respiratory muscle weakness (Pi,max < 70cmH2O)
* Persistent dyspnea on daily life (Baseline Dyspnea Index focal score <or= 8).

Exclusion Criteria:

* Inability to perform exercise tests
* Diagnosed psychiatric or cognitive disorders
* Progressive neurological or neuromuscular disorders having a major impact on exercise capacity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Dyspnea on daily life | 8 weeks
  Measured by the Baseline Dyspnea Index (BDI)

SECONDARY OUTCOMES:
Inspiratory muscle strength as measured by spirometry | 8 weeks
  Measured by Maximal Static Inspiratory Pressures (Pi,max)
Inspiratory muscle endurance as measured by a PowerBreathe device | 8 weeks
  Assessed by Endurance Respiratory Muscle Protocol (Patients will breathe against 60% of Pi,max inspiratory load until task failure)
Dyspnea on exertion | 8 weeks
  Measured by Borg score during high intensity constant load cycling exercise test
Time to exercise intolerance (Tlim) | 8 weeks
  Evaluated by high intensity constant load cycling exercise test

OTHER OUTCOMES:
Lung hyperinflation | 8 weeks
  Evaluated by serial measurements of inspiratory capacity during high intensity constant load cycling exercise test
Endothelial function as measured by non-invasive ultrasound images of the brachial artery. | 8 weeks
  Measured by ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery
Autonomic function as measured by a 10 lead ECG (MASON-LIKAR Lead electrode placement) | 8 weeks
  Measured by heart rate variability explored in the frequency domain

CONTACTS AND LOCATIONS:
Overall Officials: J Alberto Neder, MD, PhD, Study Chair — Queen's University
Locations (3):
- KU Leuven, Leuven, Belgium
- Brazil (2):
  - Universidade Federal do Rio Grande do Sul/Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No